CLINICAL TRIAL: NCT05306678
Title: Acute Effects of Breaking Prolonged Sitting on Postprandial Glycaemic Response, Incretin Hormones Secretion and Eating Behaviour in Overweight and Obese Adults
Brief Title: Breaking Sitting and Metabolic Health in Sedentary Overweight and Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yung-Chih Chen, Principal Investigator, National Taiwan Normal University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 201912HM107-
Record Dates: First submitted 2022-03-15; First posted 2022-04-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Metabolic Health; Gut Hormones; Energy Balance
Keywords: GLP-1; PYY; Breaking sitting; Energy balance; Postprandial glycaemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged sitting (Experimental): Prolonged sitting
  Interventions: Behavioral: Prolonged sitting
- Breaking sitting (Experimental): Breaking prolonged sitting
  Interventions: Behavioral: Breaking sitting

INTERVENTIONS:
Behavioral: Prolonged sitting — After consuming breakfast, participants sat on a chair for 180 min. After 180 min, lunch was provided. After finishing lunch, participants sat on a chair for another 120 min.
  Arms: Prolonged sitting
Behavioral: Breaking sitting — After consuming breakfast, participants walked 2 min on a treadmill every 20 minutes for the following 180 min. For the remainder of the time participants sat on the chair. After 180 min, lunch was provided. After finishing lunch, participants continued 2 min of walking every 20 min for the following 120 min.
  Arms: Breaking sitting

SUMMARY:
The purpose of this project is to investigate the effects of breaking up prolonged sitting on postprandial metabolic responses, gut hormones secretion and energy balance in sedentary overweight and obese adults.

DETAILED DESCRIPTION:
Two trials are included in this project - Prolonged sitting and Breaking sitting.

In the Prolonged sitting trial, after consuming breakfast, participants sat on a chair for 180 min. After 180 min, lunch was provided. After finishing lunch, participants sat on a chair for another 120 min. In the Breaking sitting trial, after consuming breakfast, participants walked 2 min on a treadmill every 20 minutes for the following 180 min. For the remainder of the time participants sat on the chair. After 180 min, lunch was provided. After finishing lunch, participants continued 2 min of walking every 20 min for the following 120 min. Blood samples were collected in a regular pattern throughout the trials. Energy balance (e.g., energy intake and spontaneous physical activity) was assessed using food diary and an accelerometer until midnight in the trial days once participants left laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Physical inactive males and females
* Aged between 20 and 45 years
* Overweight and obese healthy adults (waist circumference greater than 90 cm for males and 80 cm for females)
* Weight stable for more than 3 months (no change in weight +/- 3%)
* Non-smoker
* Able to walk comfortably on a treadmill

Exclusion Criteria:

* Personal history of/existing diabetes, cardiovascular disease, metabolic disease or dyslipidaemia
* Waist circumference < 90 cm for male and < 80 cm for female
* Taking medications that may influence lipid or carbohydrate metabolism or immune system function
* Unable to take part in exercise for any reason (e.g., injury or disability) or a positive response to any questions on the Physical Activity Readiness questionnaire (PAR-Q)

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Gut hormones responses | 320 minutes
  Changes in blood gut hormones responses (e.g., GLP-1, PYY and GIP concentrations measured in pmol/L) between trials

SECONDARY OUTCOMES:
Visual analogue scale (VAS) | 320 minutes
  Changes in VAS from 0-100 mm (e.g., appetite and mood, etc.) between trials
Energy intake | 600 minutes after leaving the labalotory
  Changes in energy intake (e.g, using a food diary to record) after leaving the laboratory until midnight
Physical activity level | 600 minutes after leaving the labalotory
  Changes in physical activity level (e.g., using an accelerometer to record) after leaving the laboratory until midnight
Lipid profile | 320 minutes
  Changes in blood lipid profile (e.g., TAG and cholesterol, etc.) between trials
Blood pressure | 320 minutes
  Changes in blood pressure (e.g., diastolic and systolic blood pressure) between trials
Computerized cognitive testing | 320 minutes
  Changes in cognitive function (e.g., accuracy and reaction time) between trials
Incremental area under curve (iAUC) for metabolic health | 320 minutes
  Changes in incremental area under curve (iAUC) for insulin and glucose between trials

CONTACTS AND LOCATIONS:
Overall Officials: Chen, PhD, Principal Investigator — National Taiwan Normal University
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No